CLINICAL TRIAL: NCT02208401
Title: A Prospective Randomised Comparison of Cold Snare Polypectomy Versus Cold Snare Pseudosuction Technique
Brief Title: Randomised Comparison of 2 Cold Snare Polypectomy Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STH17227
Record Dates: First submitted 2014-07-30; First posted 2014-08-05 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Bowel Cancer
MeSH Terms: conditions — Intestinal Neoplasms | interventions — Suction

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional cold snare polypectomy (Active Comparator): conventional cold snare polypectomy
  Interventions: Procedure: conventional cold snare polypectomy
- Cold snare polypectomy with suction (Experimental): Cold snare polypectomy with suction
  Interventions: Procedure: Cold snare polypectomy with suction

INTERVENTIONS:
Procedure: conventional cold snare polypectomy — conventional cold snare polypectomy
  Arms: conventional cold snare polypectomy
Procedure: Cold snare polypectomy with suction — Cold snare polypectomy with suction
  Arms: Cold snare polypectomy with suction

SUMMARY:
Different modalities are employed to remove small colonic polyps which potentially harbour a cancer risk. But, they can all vary in their completeness of removal, safety and the histological quality and the gold standard technique has yet to be defined. A novel suction pseudopolyp technique has been described by Patullo et al and in their prospective study, 126 polyps measuring less than 10mm flat or sessile were removed by this method with 100% complete endoscopic resection and without any immediate or delayed complications. The aim of the investigators study is to compare this technique with the standard cold snare technique. Patients attending for a routine colonoscopy and found to have polyps measuring 37mm in size will be eligible and they will be randomised to the polypectomy technique. Patient demographics and polyp characteristics will be recorded. The primary outcome measured will be the macroscopic resection rate. The secondary outcome measures are abdominal pain, tenderness, bleeding and fever.

ELIGIBILITY:
Inclusion Criteria:

* All patients with small polyps 3-7 mm in size, flat or sessile found during colonoscopy

Exclusion Criteria:

* Patients are less than 18 years old
* Pregnant
* Inadequate bowel preparation
* On anticoagulants or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Complete macroscopic polyp eradication rate | At time of polypectomy intervention
  The primary outcome for this study is the polypectomy completion rate. This will be assessed both macroscopically and histologically. The analysis for statistical difference between the 2 techniques and abdominal symptoms will be compared by the Chi2 test for categorical data.

CONTACTS AND LOCATIONS:
Overall Officials: Shawinder Johal, MBChB, PhD, MRCP, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] Din S, Ball AJ, Riley SA, Kitsanta P, Johal S. A randomized comparison of cold snare polypectomy versus a suction pseudopolyp technique. Endoscopy. 2015 Nov;47(11):1005-10. doi: 10.1055/s-0034-1392533. Epub 2015 Jul 10. PMID 26165735